CLINICAL TRIAL: NCT04743427
Title: EFFECTS OF BODY-BLADE EXERCISES ON NECK POSTURE, FUNCTION, AND MUSCLE STRENGTH IN FORWARD HEAD POSTURE
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, Nourhan Ahmed Gamal Eldin Sarhan, physical therapist at Mansheyet El Bakry General Hospital,, Cairo University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: Forward head posture treatment
Record Dates: First submitted 2021-02-03; First posted 2021-02-08 (Actual); Last update posted 2021-02-08 (Actual); Status verified 2021-01

CONDITIONS: Forward Head Posture
MeSH Terms: interventions — Exercise

STUDY DESIGN:
Intervention Model Description: Double-Blinded Randomized Controlled Trial (one investigator to make the assessment,and another investigator for application of the treatment procedures)
Who Masked: Care Provider, Investigator
Masking Description: Double (Care provider,investigator)
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- physical therapy inervention (Experimental): 1. hot pack
  2. Three active exercises
  Interventions: Other: hot pack and exercises
- Body-blade exercises in addition to physical therapy intervention (Experimental): 1. Three Body-blade exercises will be performed in random order (Two sets of, 3-minute exercise and 5-minute break, for each exercise )
  2. hot pack
  3. Three active exercises
  Interventions: Other: hot pack and exercises; Device: body blade(BB)

INTERVENTIONS:
Other: hot pack and exercises — 20-minute hot pack,and three active exercises: (a) chin tucks in supine lying with the head in contact with the floor, (b) active Standing Shoulder pull back , and (c) scapular plane shoulder elevation. (3 sets of 10 repetitions for all the 3 exercises)
Device: body blade(BB) — The Body-blade (Classic, Mad Dogg Athletics, USA), an elastic pole exercise tool with 122 cm in length, 0.68 kg, 4.3 cm in width,based on oscillatory/vibration motions that have been used in training or rehabilitation.The body blade works by rapidly changing directions at a low-frequency rhythm of approximately 4.5 Hz (cycles per second )
  Arms: Body-blade exercises in addition to physical therapy intervention

SUMMARY:
This study will be conducted to determine the effect of adding Body-blade exercises to traditional treatment on posture, scapular muscles strength, neck pain, and function in individuals with forward head posture

DETAILED DESCRIPTION:
Many studies have proposed that the Body-blade may be a more effective tool for activating the muscles employed during the training and rehabilitation of the shoulder and trunk than traditional interventions such as cuff weights and Therabands. There is few literature which studied the effect of Body-blade exercises on neck problems. So there is insufficient evidence for their effectiveness on improving forward head posture.

ELIGIBILITY:
Inclusion Criteria :

1. Participants with FHP of both genders
2. Age range from 20-40 years
3. craniovertebral angle (CVA) less than 52 degrees

Exclusion Criteria :

1. Patients with a previous diagnosis of a musculoskeletal system disease over the last 6 months,
2. severely unstable spine
3. osteoporosis
4. vascular disease
5. cervical or shoulder neurological movement disorder

Ages: 20 Years to 40 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 42 (Estimated)
Dates: Start 2020-12-30 (Actual); Primary Completion 2021-04 (Estimated); Study Completion 2021-08 (Estimated)

PRIMARY OUTCOMES:
cranio vertebral angle using the Autocad | 5 minutes
  It is defined as the angle formed from a horizontal line passing through the C7 spinous process and a line passing through the tragus of the ear

SECONDARY OUTCOMES:
pain using visual Analogue Scale (VAS) | 5 minutes
  VAS is a self-reported scale consisting of a horizontal or vertical line, usually 10 centimeters long (100 mm) anchored at the extremes by two verbal descriptors referring to the pain status
Neck function using the Neck Disability Index | 5 minutes
  The participants will be informed with the questionnaire10-items: pain intensity, personal care, lifting, work, headaches, concentration, sleeping, driving, reading, and recreation. and will be asked to fill the response to each item which is rated on a 6-point scale from 0 (no disability) to 5 (complete disability).The higher the final score the more severe the functional disability. Scores were divided into 0- 4 points for no disability, 5-14 points for mild disability, 15-24 points for moderate disability, 25-34 points for severe disability, and 35 or higher for complete disability
Scapular muscles strength using Hand Held Dynamometer | 10 minutes
  the participants will be positioned in different positions according to the muscle to be measured .

CONTACTS AND LOCATIONS:
Locations (1):
- Mansheyet El Bakry General Hospital, Cairo, Egypt

REFERENCES:
- [Background] Sheikhhoseini R, Shahrbanian S, Sayyadi P, O'Sullivan K. Effectiveness of Therapeutic Exercise on Forward Head Posture: A Systematic Review and Meta-analysis. J Manipulative Physiol Ther. 2018 Jul-Aug;41(6):530-539. doi: 10.1016/j.jmpt.2018.02.002. Epub 2018 Aug 11. PMID 30107937
- [Background] Lister JL, Del Rossi G, Ma F, Stoutenberg M, Adams JB, Tobkin S, Signorile JF. Scapular stabilizer activity during Bodyblade, cuff weights, and Thera-Band use. J Sport Rehabil. 2007 Feb;16(1):50-67. doi: 10.1123/jsr.16.1.50. PMID 17699887